CLINICAL TRIAL: NCT03522597
Title: Maternal Metabolism, Breast Milk Composition, and Infant Outcomes: The 4M Project
Brief Title: Metabolism, Breastmilk, and Microbiome
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Oklahoma (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: OBGYN-2018-26409; R01HD080444 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-05-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Diabetes, Gestational
Keywords: Obesity; Gestational Diabetes; Breast Milk; Microbiome; Infant Growth
MeSH Terms: conditions — Obesity; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal serum and breast milk, infant feces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal weight: Normal weight (BMI) women and their infants
- Obese: Obese (BMI) women and their infants
- Diabetic: Women with gestational diabetes and their infants

SUMMARY:
The objective of this pilot study is to compare breast milk composition in mothers of three different metabolic states (normal weight, obese, and gestational diabetic) and to determine the extent to which breastmilk components are transmitted to the infant gut and are associated with the anthropometric and body composition changes in their infants during the first 6 months of life. It is hypothesized that 1) different maternal metabolic states will be associated with differences in breastmilk microbial communities and breastmilk biochemical features, 2) differences in these breastmilk biomarkers will be transmitted to infants and 3) breastmilk microbial and metabolic features will be associated with infant growth outcomes.

DETAILED DESCRIPTION:
The incidence of both obesity and diabetes are on a staggering rise. Many studies suggest that by 2030, 40-50% of the population will be obese. The prevalence of gestational diabetes (GDM) is also increasing, and was recently reported to be 9%. GDM increases risk of obesity and impaired glucose tolerance in their children, but the mechanisms by which this occurs are not well defined.

The benefits of breastfeeding are numerous, including protection from sudden infant death and infection, positive cognitive outcomes, reduced prematurity complications, and decreased risk of cancer, as well as some evidence of protection against child obesity. One area that has yet to be thoroughly explored is whether there are differences in breast milk composition in women with diabetes as compared to non-diabetic women after adjusting for obesity and other diabetes co-morbidities, and how these differences could affect infant metabolic health and body composition. Experimental studies argue strongly for a causal relationship of the gut microbiome to the risk of obesity and diabetes. Breast milk strongly shapes the gut microbiome, as it contains unique oligosaccharides as well as hormones and immunologic factors that cultivate the growth of specific microbiota in the infant gut. Indeed over 90% of early infant fecal bacteria are Bifidobacteria, where in most formula-fed infants Bifidobacteria are non-detectable, which has been linked to the rapid growth and greater adiposity in formula-fed versus breastmilk-fed infants. Given that most pregnant women in the United States are now either overweight, obese, or diabetic, our study has high public health significance in that it seeks to understand how maternal metabolic factors such as these hinder the development of a healthy gut microbiome during the critical period of infancy.

In this study, the following study questions will be examined:1) does maternal metabolic state relate to the milk microbiome (bacterial and fungal diversity and abundance relationships, and microbiome function) and how they are transmitted to the infant gut? 2) does maternal metabolic state relate to the concentration of appetite and growth-regulating hormones and cytokines present in breast milk?; 3) are maternal serum concentrations of hormones and milk microbiomes associated with each other?; and 4) are milk hormones and/or milk microbiomes related to infant growth and body composition in the first 6 months of life?

Amplicon-based and deep (shotgun) metagenomic sequencing will be utilized to characterize species and strain level characteristics of maternal milk and infant fecal microbiomes. ELISA assays will be used to quantify adipose-tissue derived hormones (leptin, adiponectin) and immune factors (CRP, IL-6, TNF-α) as well as insulin/growth axis hormones (insulin, IGF-1, IGFBP-3) in breast milk. Infant body composition will be assessed using air displacement plethysmography and dual energy x-ray absorptiometry.

The above work will involve new recruitment enrollment, and pregnancy data collection from 50 diabetic mothers recruited through the Maternal Fetal Medicine and Women's Health Specialists at M Health. The pregnant non-diabetic (normal weight and obese) woman cohorts (and their infants and samples) for this study already exist as part of Clinical Trial NCT03301753 (Maternal Obesity, Breast Milk Composition, and Infant Growth (MILK) study), which is currently in the sample collection phase. The current study will form the first comprehensive comparison of multiple aspects of breastmilk composition in women with pregnancy diabetes as compared to non-diabetic women.

ELIGIBILITY:
Inclusion Criteria:

(For new enrollment of 50 pregnant women with gestational diabetes and their infants. Enrollment of normal weight and obese cohort comparators already accomplished under ClinicalTrial NCT03301753):

1. Pregnant women
2. age 21-45 at time of delivery
3. report during enrollment procedures that they have social support for and intention to exclusively breastfeed for at least 3 months (breastfeeding intentions are known to be correlated with actual behavior), and if parity >1, that they successfully breastfed after a previous pregnancy for at least 3 months
4. singleton pregnancy
5. known gestational diabetes Definition of Gestational Diabetes: 1) an elevated glucose challenge test >200 mg/dL or 2) two abnormal values on the glucose tolerance test according to Carpenter-Coustan criteria.

Exclusion Criteria:

1. alcohol consumption >1 drink per week during pregnancy/lactation
2. tobacco consumption during pregnancy/lactation,
3. inability to speak/understand English
4. known congenital metabolic, endocrine disease, or congenital illness affecting infant feeding
5. planned delivery at a site other than the University of Minnesota Medical Center- West Bank campus.
6. preexisting diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: (for new enrollment of 50 pregnant women with gestational diabetes and their infants. Enrollment of normal weight and obese cohort comparators already accomplished under ClinicalTrial NCT03301753) Recruitment of women with gestational diabetes will be conducted at the University of Minnesota Medical Center (UMMC) Department of Obstetrics, Gynecology, and Women's Health, Division of Maternal Fetal Medicine and Women's Health Specialists Clinics (Minneapolis, MN) during an antenatal clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 2050 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Breastmilk and infant microbiomes | 1, 3, and 6 months postpartum
  Change in the diversity and abundance of breast milk and infant gut bacterial and fungal species and strains, and functional microbiome profiles

SECONDARY OUTCOMES:
Hormones in breastmilk | 1 and 3 months postpartum
  Change in breastmilk concentrations of appetite and growth regulating hormones (leptin, insulin, adiponectin) and proteins (IGF-1, IGFBP3, CRP, IL-6) from milk.
Hormones and cytokines in maternal serum | At time of delivery (time 0)
  Maternal serum concentrations of appetite and growth regulating hormones (leptin, insulin, adiponectin) and proteins (IGF-1, IGFBP3, CRP, IL-6), and cytokines.
Hormones and cytokines in infant serum | At time of delivery (time 0) and 6 months postpartum
  Change in the concentrations of appetite and growth regulating hormones (leptin, insulin, adiponectin) and proteins (IGF-1, IGFBP3, CRP, IL-6), and cytokines from birth to age 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Gale, M.D., Principal Investigator — University of Minnesota; Ellen W Demerath, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No